CLINICAL TRIAL: NCT01494090
Title: Efficacy and Safety of Rosuvastatin in the Prevention of Arterial and Venous Vascular Events and Mortality After Hip Fracture: A Multicenter Randomised, Double-blinded, Placebo Controlled Trial.
Brief Title: Statin in Hip Fracture
Acronym: STAFF
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Decision of the Steering Committee. Recruitment more difficult and slower than expected.
Sponsor: University Hospital, Brest (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RB 10-094 STAFF
Record Dates: First submitted 2011-12-15; First posted 2011-12-16 (Estimated); Last update posted 2012-09-20 (Estimated); Status verified 2012-09

CONDITIONS: Hip Fracture
Keywords: Venous thromboembolism; Hip fracture; Cardiovascular events; Statin
MeSH Terms: conditions — Hip Fractures; Venous Thromboembolism | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rosuvastatin (Active Comparator)
  Interventions: Drug: Rosuvastatin
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rosuvastatin — 5 or 20 mg per day during 6 months
  Arms: Rosuvastatin
Drug: Placebo — 5 or 20 mg per day during 6 months
  Arms: placebo

SUMMARY:
Statins (or HMG-CoA reductase inhibitors) have largely proven their efficacy in the primary and secondary prevention of cardiovascular events. Many clinical and experimental studies support also a potential beneficial effect of statin therapy on venous thromboembolism (VTE). Patients with hip fracture are at high risk of VTE and cardiovascular events.

The aim of this study is to evaluate the efficacy and the tolerance of a statin (rosuvastatin) in hip fracture surgery on the occurrence of venous and atherothrombotic events and the global mortality at six months.

Subjects aged 60 years or over who are scheduled to undergo surgery for fracture of the upper portion of the femur (hip fracture) are eligible to participate to this multicentre, randomized, double-blind placebo controlled trial. They will receive either rosuvastatin (5 or 20 mg) or placebo for 6 months. The primary efficacy outcome is the incidence of an adjudicated composite of non fatal VTE, acute coronary syndrome, non fatal stroke, other acute ischemic arterial event, or all-cause death.

Assuming a endpoint frequency of 20% in the control group, we calculated that 1200 patients will be required for the study to have 80% power to detect a 30% reduction in the relative risk with rosuvastatin (with a two-sided alpha level of 5%).

The investigators assumed that rosuvastatin could have a positive benefit-risk ratio in patients undergoing orthopaedic surgery for hip fracture, by reducing vascular events and global mortality at six months.

ELIGIBILITY:
Inclusion Criteria:

* 60 years old or older.
* fracture of the femoral neck or of the trochanteric mass
* undergoing surgery within 5 days for this fracture
* Signed written informed consent

Exclusion Criteria:

* contraindication to rosuvastatin:
* active liver disease including unexplained and prolonged elevations of serum transaminases and any increase of serum transaminases beyond 3 times the upper limit of normal
* severe renal impairment (creatinine clearance calculated by the formula MDRD <30 ml / min)
* myopathy
* use of cyclosporine
* statin therapy ongoing at the admission for fracture
* curative anticoagulant therapy ongoing at the admission and expected to be maintained after the intervention
* Patients considered by the investigator to be unable to participate to the study
* Refuse to participate

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2011-08; Primary Completion 2012-03 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Occurence of Arterial and Venous Vascular Events and Mortality | 6 months
  * Nonfatal symptomatic thromboembolic venous desease
  * Acute coronary syndrome
  * Nonfatal ischemic stroke or transient ischemic attack
  * Acute peripheral arterial ischemia
  * Deaths from all causes

CONTACTS AND LOCATIONS:
Overall Officials: Dominique MOTTIER, Principal Investigator — University Hospital, Brest
Locations (6):
- France (6):
  - Brest, University Hospital, Brest
  - Caen, University Hospital, Caen
  - Grenoble, University Hospital, Grenoble
  - APHP - Cochin Hospital, Paris
  - Quimper Hospital, Quimper
  - St-Etienne, University Hospital, Saint-Etienne